CLINICAL TRIAL: NCT05846295
Title: Online Education Module (ESTIMATE: Estimating Polyp Size With Snare Tool to Improve Measurement Accuracy for Trainee Education) to Accurately Classify Polyp Size
Brief Title: Online Education Module to Accurately Classify Polyp Size
Acronym: ESTIMATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of California, San Francisco (Other); Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: 20-1413
Record Dates: First submitted 2023-03-28; First posted 2023-05-06 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Polyp; Colonic Neoplasms
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is an educational intervention study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigators will be blinded regarding which participants are randomized to which arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): No video tutorial, no feedback
- Feedback (Active Comparator): Feedback only
  Interventions: Other: ESTIMATE
- Video (Active Comparator): Video tutorial only
  Interventions: Other: ESTIMATE
- Video + Feedback (Experimental): VIdeo tutorial and feedback
  Interventions: Other: ESTIMATE

INTERVENTIONS:
Other: ESTIMATE — An online educational module consisting of a video tutorial and feedback during a questionnaire
  Arms: Feedback; Video; Video + Feedback

SUMMARY:
Investigators developed an online educational module (ESTIMATE) to teach Gastroenterology (GI) trainees how to estimate polyp size using a snare. Key components include video instruction and real-time feedback incorporated over a 40-item polyp size assessment test. Trainees from GI fellowship programs will be randomized to one of four groups: control (no video, no feedback), video-only, feedback-only, and video + feedback. Participants will classify polyps into one of three size categories:- diminutive (1-5 mm), small (6-9 mm), and large (≥10 mm). Primary outcome is accuracy of polyp size classification [diminutive (1-5 mm), small (6-9 mm), and large (≥10 mm)]. Secondary outcomes include accuracy of exact polyp size (in mm), cumulative accuracy (to plot learning curves), confidence level of polyp size classification, and directionality of inaccuracy (polyp size overestimation vs underestimation).

DETAILED DESCRIPTION:
Study Design This is a prospective, multicenter educational randomized controlled trial. Trainees from five Accreditation Council for Graduate Medical Education (ACGME)-accredited GI fellowship training programs in the US will be invited to participate.

Study Materials (ESTIMATE Online Educational Module) The Estimating Polyp Size with Snare Tool to Improve Measurement Accuracy for Trainee Education (ESTIMATE) online educational module was developed by the study team over an 11-month development phase from September 2020 - August 2021. ESTIMATE is a user-friendly, interactive, web-based teaching module consisting of two main educational components: (1) video instruction and (2) real-time feedback during a polyp size assessment test. Video instruction is provided in a five-minute didactic clip that narrates the importance of accurate polyp size classification and demonstrates proper technique for positioning the snare to estimate polyp size. Examples of both correct and incorrect technique are provided. Several case examples, with opportunity for trainee interaction and response, are also included.

The polyp size assessment test includes 40 polyp sizing questions. Each question contains a still image of a polyp with an adjacent snare and asks participants to correctly identify the polyp's size into one of the following clinically relevant size categories: diminutive (1-5 mm), small (6-9 mm), and large (≥10 mm), as well as the exact polyp size in mm. Participants are also asked to provide their confidence level (high or low) with each response. High confidence is defined as a sufficient level of certainty in polyp size to commit to a surveillance interval recommendation based on the response. Low confidence is defined as an insufficient level of certainty in polyp size to commit to a surveillance interval recommendation based on the response.

Real-time feedback on correct polyp size is provided immediately after a response is submitted in the form of a series of images with overlying graphics that demonstrate polyp size relative to the adjacent snare with a final image of the resected polyp affixed to a cork board and ruler. Investigators used measurement of the immediate post-resection, pre-formalin fixation polyp affixed to a cork board with an adjacent ruler to determine correct size. The feedback image deck will be provided in continuous fashion after each response as participants progress through the test.

Randomization In order to assess the impact of the key educational components of our module (video instruction and feedback), participants will be randomized in REDCap to one of four study groups: control, video-only, feedback-only, or video + feedback. The control group will complete the 40-item polyp size assessment test without receiving any video instruction or feedback. The video-only group will watch the video instructional clip and then completed the assessment, but will not receive any feedback after each question. The feedback-only group will receive feedback after each question, but will not watch the video. Lastly, the video + feedback group will receive both video instruction and feedback as they complete the assessment.

Data Collection and Reporting System All data will be collected and managed using Research Electronic Data capture (REDCap).

Statistical Analysis & Sample Size Considerations Bivariable analyses will be performed to identify potential differences between groups. Binomial regressions will be conducted to detect differences between the control and intervention groups in accuracy of polyp size by size classification and exact size in mm. Generalized linear mixed models will be used to assess differences in confidence while accounting for multiple responses within each participant. Models will be evaluated using a type I error rate of 0.05. Analyses will be conducted using R version 4.1.1. In order to achieve 80% power to detect a 20% difference between the three intervention groups and the control group, we will need to enroll twelve trainees within each group (48 total).

ELIGIBILITY:
Inclusion Criteria:

* GI trainees who have never received formal training in, nor had participated in a research study on, polyp sizing
* Informed consent

Exclusion Criteria:

* Those who do not complete the educational module during the allotted time

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2024-12-28 (Estimated)

PRIMARY OUTCOMES:
Participant entered rate of accurate polyp size classification into diminutive (1-5 mm), small (6-9 mm), or large (≥10 mm) category on 40 question polyp sizing test. | through study completion, estimated 1 year
  The gold standard polyp size for the polyp images on the polyp sizing test was determined by affixing the polyp to a cork board post-procedure and measuring it with an adjacent ruler. The actual polyp size was determined by meauring it against the adjacent ruler. Polyps 1-5 mm were categorized as diminutive, polyps 6-9 mm were categorized as small and polyps ≥10 mm were categorized as large.
  Participants completed a 40 item polyp sizing test where participants designated the polyp as either dimunitive (1-5mm), small (6-9mm) or large (≥10mm). The primary outcome was the rate that each participant correctly designated polyp size categories based on the gold standard.

SECONDARY OUTCOMES:
Participant entered rate of accurate polyp size by millimeter on 40 question polyp sizing test. | through study completion, estimated 1 year
  Participant rate of accurate polyp size by millimeter (1mm, 2mm, 3mm, 4mm, 5mm, 6mm, 7mm, 8mm, 9mm, 10mm, 11mm, 12mm, 13mm, 14mm, 15mm, 16mm, 17mm, 18mm, 19mm, 20mm, etc) on 40 question polyp sizing test.
Cumulative accuracy of polyp size category classification as participants progress through the 40 item polyp sizing test | through study completion, estimated 1 year
  Cumulative accuracy of polyp size category classification as participants progress through the 40 item polyp sizing test
Participant report of categorical high versus low confidence on each response of the 40 item polyp sizing test | through study completion, estimated 1 year
  self-reported high vs low confidence of each polyp characterization. High confidence is defined as sufficient self-assessed confidence that participant can make a post-polypectomy surveillance interval recommendation based on their designation. This is categorical selection of "high" vs "low"
Proportion of participant responses that underestimate actual polyp size category versus overestimate actual polyp size category on the 40-question polyp sizing test. | through study completion, estimated 1 year
  Proportion of responses that underestimate actual polyp size category (a small or large polyp categorized as diminutive or a large polyp categorized as small) versus overestimate actual polyp size category (a diminutive or small polyp characterized as large or a diminutive polyp characterized as small).

CONTACTS AND LOCATIONS:
Overall Officials: Swati G Patel, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta S, Lieberman D, Anderson JC, Burke CA, Dominitz JA, Kaltenbach T, Robertson DJ, Shaukat A, Syngal S, Rex DK. Recommendations for Follow-Up After Colonoscopy and Polypectomy: A Consensus Update by the US Multi-Society Task Force on Colorectal Cancer. Am J Gastroenterol. 2020 Mar;115(3):415-434. doi: 10.14309/ajg.0000000000000544. No abstract available. PMID 32039982
- [Background] Gopalswamy N, Shenoy VN, Choudhry U, Markert RJ, Peace N, Bhutani MS, Barde CJ. Is in vivo measurement of size of polyps during colonoscopy accurate? Gastrointest Endosc. 1997 Dec;46(6):497-502. doi: 10.1016/s0016-5107(97)70003-8. PMID 9434215
- [Background] Chaptini L, Chaaya A, Depalma F, Hunter K, Peikin S, Laine L. Variation in polyp size estimation among endoscopists and impact on surveillance intervals. Gastrointest Endosc. 2014 Oct;80(4):652-659. doi: 10.1016/j.gie.2014.01.053. Epub 2014 Mar 27. PMID 24679658
- [Background] Utsumi T, Horimatsu T, Seno H. Measurement bias of colorectal polyp size: Analysis of the Japan Endoscopy Database. Dig Endosc. 2019 Sep;31(5):589. doi: 10.1111/den.13447. Epub 2019 Jun 13. No abstract available. PMID 31120583
- [Background] Kaltenbach T, Anderson JC, Burke CA, Dominitz JA, Gupta S, Lieberman D, Robertson DJ, Shaukat A, Syngal S, Rex DK. Endoscopic Removal of Colorectal Lesions-Recommendations by the US Multi-Society Task Force on Colorectal Cancer. Gastrointest Endosc. 2020 Mar;91(3):486-519. doi: 10.1016/j.gie.2020.01.029. Epub 2020 Feb 14. No abstract available. PMID 32067745
- [Background] Patel SG, May FP, Anderson JC, Burke CA, Dominitz JA, Gross SA, Jacobson BC, Shaukat A, Robertson DJ. Updates on Age to Start and Stop Colorectal Cancer Screening: Recommendations From the U.S. Multi-Society Task Force on Colorectal Cancer. Am J Gastroenterol. 2022 Jan 1;117(1):57-69. doi: 10.14309/ajg.0000000000001548. PMID 34962727
- [Background] Patel SG, Rastogi A, Austin G, Hall M, Siller BA, Berman K, Yen R, Bansal A, Ahnen DJ, Wani S. Gastroenterology trainees can easily learn histologic characterization of diminutive colorectal polyps with narrow band imaging. Clin Gastroenterol Hepatol. 2013 Aug;11(8):997-1003.e1. doi: 10.1016/j.cgh.2013.02.020. Epub 2013 Mar 1. PMID 23466714